CLINICAL TRIAL: NCT02937675
Title: A Phase 1-2 Dose-Escalation and Cohort-Expansion Study of Oral Tomivosertib (eFT-508) in Subjects With Hematological Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: patient recruitment
Sponsor: Effector Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eFT508-0002
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: small molecule inhibitor of protein translation; immunomodulator; phase 1 dose escalation
MeSH Terms: conditions — Lymphoma | interventions — tomivosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tomivosertib (eFT-508) Escalation Cohort (Experimental): This portion of the study will evaluate the safety and pharmacology of a range of Tomivosertib (eFT-508) doses administered daily in subjects with previously treated lymphomas
  Interventions: Drug: Tomivosertib (eFT-508)
- Tomivosertib (eFT-508) Expansion Cohort (Experimental): This portion of the study provides cohort expansion to further explore the safety, pharmacology, and clinical activity of a single dose level of Tomivosertib (eFT-508) monotherapy in subjects with specific previously treated lymphomas
  Interventions: Drug: Tomivosertib (eFT-508)

INTERVENTIONS:
Drug: Tomivosertib (eFT-508) — eFT508

SUMMARY:
This clinical trial is a Phase 1-2, open-label, sequential-group, dose-escalation and cohort-expansion study evaluating the safety, pharmacokinetics, pharmacodynamics, and antitumor activity of Tomivosertib (eFT-508). The study will evaluate oral daily administration of Tomivosertib (eFT-508). Treatment and study subject evaluation will be performed in 21-day cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
2. Presence of an active hematological malignancy.
3. Presence of measurable disease.
4. Hematological malignancy has been previously treated, has relapsed after or progressed during prior therapy, and has limited potential for benefit from currently available therapy including hematopoietic stem cell transplantation.
5. At least 2 weeks post any treatments/therapies at the time of first dose.
6. Adequate bone marrow function.
7. Adequate hepatic function.
8. Adequate renal function.
9. Normal coagulation panel.
10. Negative antiviral serology.
11. Willingness to use effective contraception.

Exclusion Criteria:

1. Central nervous system malignancy
2. Gastrointestinal disease
3. Significant cardiovascular disease
4. Significant ECG abnormalities.
5. Ongoing risk for bleeding due to active peptic ulcer disease, bleeding diathesis or requirement for systemic anticoagulation
6. Ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections)
7. Pregnancy or breastfeeding.
8. Major surgery within 4 weeks before the start of study therapy.
9. Ongoing immunosuppressive therapy, including systemic or enteric corticosteroids
10. Use of drugs that could prolong the QT interval within 7 days before the start of study therapy.
11. Use of drugs that might pose a risk of a drug-drug interaction within 2-7 days before the start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and/or Recommended Dose within the tested Tomivosertib (eFT-508) dose range | up to one year
Overall Response Rate | up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Barton, MD, Study Director — CMO
Locations (10):
- United States (10):
  - Samuel Oschin comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Florida Cancer Specialist, Sarasota, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester, Rochester, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No